CLINICAL TRIAL: NCT00490100
Title: Treatment for Growth Failure in Patients With X-Linked Severe Combined Immunodeficiency (XSCID): A Phase 2 Study Assessing Safety and Clinical Response to Treatment With Insulin-like Growth Factor-1 (IGF-1)
Brief Title: Treatment for Growth Failure in Patients With X-Linked Severe Combined Immunodeficiency: Phase 2 Study of Insulin-Like Growth Factor-1
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Insufficient patient participation
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070171; 07-I-0171
Record Dates: First submitted 2007-06-21; First posted 2007-06-22 (Estimated); Results first posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2014-03

CONDITIONS: Growth Failure; X-linked Severe Combined Immunodeficiency (XSCID); Growth Hormone Resistence
Keywords: X-Linked Severe Combined Immune Deficiency (XSCID); Growth Hormone; Insulin-Like Growth Factor 1 (IGF)-1; Bone Age; Growth Failure; XSCID; X-Linked Severe Combined Immunodeficiency
MeSH Terms: conditions — Failure to Thrive; X-Linked Combined Immunodeficiency Diseases | interventions — mecasermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Treatment
  Interventions: Drug: Increlex

INTERVENTIONS:
Drug: Increlex

SUMMARY:
This study will evaluate the safety and effectiveness of insulin-like growth factor-1 (IGF-1) to treat patients with X-linked severe combined immunodeficiency (XSCID). Those who have XSCID lack white blood cells that protect their bodies from invasion by all types of germs. IGF-1 is the main hormone responsible for the body's growth and metabolism. As a medication, IGF-1 is Increlex[(Trademark)] (mecasermin),

Patients ages 2 to 20 who have not yet begun puberty, have a diagnosis of XSCID, and are shorter than the 3rd percentile for their age may be eligible for this study. This study will last about 3 years, and patients' visits will be scheduled at 3-month intervals. Patients will have a physical history and exam, X-rays, electrocardiogram, blood tests, and body measurements.

Patients will take estradiol orally for 2 days, to help avoid false results of growth hormone (GH) levels in blood samples. Then provocation testing is done, with two tests back to back. It determines blood levels of GH and the body's response to testing with drugs called arginine and clonidine. Patients are admitted to the pediatric inpatient unit and will have an intravenous (IV) line placed in the arm. Arginine is given by IV over 30 minutes, and blood samples are taken. Right after arginine testing, the clonidine tablet is given. The IGF-1 generation test is then done to see if the body makes IGF-1 as a product in response to injections of GH for 5 consecutive days. This test does not require that patients are inpatients, but after Day 8, patients must be admitted to the pediatric unit to have blood sampling, start Increlex injections, and start close monitoring of blood sugar levels. They will learn how to do a self-injection and follow other advice. They will complete records about the injection site, symptoms, and side effects-keeping records for at least the first 2 days after going home, with each dose change, and as needed. Patients stick their fingertip and place a small drop of blood on a blood sugar monitoring strip. The strip is put into a glucometer-a small hand-held device to measure the blood sugar level. Patients will be instructed to always have a source of sugar available in case blood sugar is too low.

...

DETAILED DESCRIPTION:
This is a Phase 2 protocol evaluating the safety and efficacy of standard dose insulin-like growth factor-1 (IGF-1) for the treatment of growth failure in patients diagnosed with X-linked severe combined immunodeficiency (XSCID). This condition is a fatal inherited immunodeficiency caused by defects in the common cytokine receptor gamma chain (gc), a subunit shared by many cytokine receptors. The common gamma subunit signals through the Janus kinase/signal transducers and activators of transcription (JAK/STAT) pathway, a complex intracellular signaling pathway used by many cytokines and growth factors, including growth hormone (GH). Studies have suggested that the gc defect may result in hyporesponsiveness to GH. This is supported by a report of GH hyporesponsiveness in an XSCID child that was successfully ameliorated following immune reconstitution using bone marrow transplantation (BMT). Haplo-identical BMTs for XSCID children often achieve only partial immune reconstitution, and many BMT recipients experience ongoing problems with growth failure, achieving heights well below 2 standard deviations for their chronological age. It is possible that in these partially corrected conditions, administration of IGF-1, a substance the body produces downstream in response to GH, may achieve an improved growth response.

This study proposes to evaluate the safety and efficacy of Increlex(Trademark) (recombinant human IGF-1) for the treatment of patients with XSCID who have growth failure (children with heights less than 3rd percentile for age). Increlex(Trademark) is a Food and Drug Administration-approved drug for treatment of growth hormone non-responsiveness in the general population of children with growth hormone hyporesponsiveness or primary IGF-1 deficiencies. The scientific objectives are to determine safety and to assess the efficacy of using subcutaneous IGF-1 in XSCID patients with growth failure. The long-term goal of this study is to establish improved treatment regimens for growth failure in children with XSCID.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants Must:

* Have a diagnosis of XSCID
* Be between 2 years to 20 years old and have not completed puberty
* Consent to permit blood and/or tissue samples for storage
* Demonstrate short stature: height below the 3 rd percentile for chronological age
* Have a primary care physician at home
* Demonstrate growth failure, defined as growth velocity (measured as linear growth) that is less than 5% to 10% of that expected for children of the same age group, over the past 12 months
* Willingness to remain hospitalized for several days
* Provide evidence of serum IGF-1 level performed within the preceding 6 months and the results fall below normal limits for age

EXCLUSION CRITERIA:

Participants Must NOT:

* Have fusion of epiphyseal plates
* Demonstrate any history of anaphylactic reaction or hypersensitivity to mecasermin or any component of the drug's formulation
* Have any active or suspected neoplasia
* Demonstrate signs of intracranial hypertension as evidenced by papilledema upon examination by fundoscopy
* Have any condition that, in the investigator's opinion, places the patient at undue risk by participating in the study
* Be unwilling to undergo testing or procedures associated with this protocol

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2007-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suk S De Ravin, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Buckley RH, Schiff RI, Schiff SE, Markert ML, Williams LW, Harville TO, Roberts JL, Puck JM. Human severe combined immunodeficiency: genetic, phenotypic, and functional diversity in one hundred eight infants. J Pediatr. 1997 Mar;130(3):378-87. doi: 10.1016/s0022-3476(97)70199-9. PMID 9063412
- [Background] Puck JM, Pepper AE, Henthorn PS, Candotti F, Isakov J, Whitwam T, Conley ME, Fischer RE, Rosenblatt HM, Small TN, Buckley RH. Mutation analysis of IL2RG in human X-linked severe combined immunodeficiency. Blood. 1997 Mar 15;89(6):1968-77. PMID 9058718
- [Background] Leonard WJ, Shores EW, Love PE. Role of the common cytokine receptor gamma chain in cytokine signaling and lymphoid development. Immunol Rev. 1995 Dec;148:97-114. doi: 10.1111/j.1600-065x.1995.tb00095.x. PMID 8825284
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-I-0171.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Participants are young males with X-linked severe combined immunodeficiency complicated by growth failure. The participants will receive Insulin-like Growth Facor (Increlex) twice a day for up to 2 years.
Period: Overall Study
Arm/Group | Treatment
Started | 6
Completed | 3
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety of Study Drug
Description: Rates of adverse events related to study drug
Time Frame: 1 year
Measure: Number; unit: participants
Groups:
- Treatment: XSCID patients with growth failre treated with Increlex, recombinant human IGF-1.
  Increlex
Arm/Group | Treatment
Number analyzed (Participants) | 3
participants | 0

2. Primary Outcome: Change in Growth Rate on Study Drug
Description: Growth rate on intervention is compared with growth rate before intervention for each participant.
Time Frame: During intervention, up to 2 years
Population: Only participants who completed study
Measure: Median (Full Range); unit: cm/year
Arm/Group | Treatment
Number analyzed (Participants) | 3
cm/year | 5.2 [1.2 to 8.6]

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=6)
Diarrhea (clostridium diff) (Gastrointestinal disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Lung infection (Infections and infestations) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Due to limited subject participation, there is insufficient complete data to generate meaningful statistics for the outcome measures. Instead, this data will be reported as a case series.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes